CLINICAL TRIAL: NCT06106919
Title: PFENDO : Ovarian Blockade During Fertility Preservation in Patients With Endometriosis: a Retrospective Non-inferiority Comparative Study
Brief Title: Ovarian Blockade During Fertility Preservation in Patients With Endometriosis
Acronym: PFENDO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2023/SH-01; 2023-A02214-41 (Other: ANSM)
Record Dates: First submitted 2023-10-20; First posted 2023-10-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- dienogest
  Interventions: Other: surveys (Fertiqol and WHOQOL-BREF)
- GnRH agonist
  Interventions: Other: surveys (Fertiqol and WHOQOL-BREF)
- GnRH antagonist
  Interventions: Other: surveys (Fertiqol and WHOQOL-BREF)

INTERVENTIONS:
Other: surveys (Fertiqol and WHOQOL-BREF) — surveys (Fertiqol and WHOQOL-BREF)

SUMMARY:
The aim of the study is to demonstrate the non-inferiority of dienogest on the number of mature oocytes collected compared with "conventional" ovarian stimulation protocols (using a GnRH agonist or antagonist), in patients with endometriosis in a fertility preservation context.

DETAILED DESCRIPTION:
Endometriosis is a common pathology affecting 1 in 10 women of childbearing age, and is responsible for around 40% of infertility cases.

The impact of endometriosis on fertility has now been clearly demonstrated, making it a medical indication for fertility preservation.

Today, dienogest is a key element in the therapeutic arsenal, helping to alleviate painful symptoms, reduce endometriosis lesions and improve patients' quality of life.

By creating a hypo-oestrogenic and hyperprogestogenic climate, dienogest at a daily dose of 2mg not only atrophies the endometrial tissue of endometriotic lesions, but also inhibits ovulation, enabling it to be used as an adjuvant treatment to ovarian stimulation.

There are currently 3 protocols commonly used during ovarian stimulation for oocyte self-preservation: the antagonist protocol (using a GnRH antagonist), the agonist protocol (using a GnRH agonist) and the PPOS protocol (using a progestin, which may be dienogest). In patients undergoing long-term dienogest therapy, the first 2 protocols require discontinuation of background treatment, which entails a risk of recurrence of symptoms and progression of endometriosis lesions, unlike the PPOS protocol, which allows dienogest treatment to be continued during stimulation.

A few studies have looked at progestin blockade of ovulation during ovarian stimulation and found no negative impact on the number of oocytes collected, compared with commonly used protocols (antagonist or agonist protocol). However, these studies do not concern blocking with dienogest, a progestin whose use has recently been extended due to the generic drug's marketing authorization obtained in 2019.

Ovarian stimulation with dienogest has therefore received very little attention in the literature. The only study on this subject is a prospective study comparing dydrogesterone and dienogest during ovarian stimulation for IVF. The number of mature oocytes collected was significantly lower in the dienogest group, but the 2 groups were not comparable, particularly in terms of AMH and CFA, which were significantly lower in the dienogest group, making the results difficult to interpret.

Further studies therefore seem necessary to investigate the impact of dienogest blockade on ovarian response, given the benefits brought by this treatment in terms of ease of use and clinical tolerance in patients with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 42 inclusive
* Patient with endometriosis
* Patient who has undergone at least one cycle of ovarian stimulation for fertility preservation between June 2022 and September 2023 inclusive, using one of the protocols studied:

GnRH agonist GnRH antagonist Dienogest

Exclusion Criteria:

-Non-medical or medical fertility preservation excluding endometriosis

Ages: 18 Years to 42 Years | Sex: Female
Age Groups: Adult
Study Population: Women of childbearing age with endometriosis who have undergone at least one cycle of ovarian stimulation for fertility preservation between June 2022 and September 2023.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes collected by ovarian puncture | through study completion, an average of 15 days
  Number of mature oocytes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calero M, Robert J, Ranisavljevic N, Petit E, Montagut M, Lesourd F, Chevalier N, Huberlant S. Fertility preservation in women with endometriosis: A retrospective non-Inferiority study comparing Dienogest in the PPOS protocol to antagonist and agonist protocols. J Gynecol Obstet Hum Reprod. 2025 Jun;54(6):102950. doi: 10.1016/j.jogoh.2025.102950. Epub 2025 Apr 3. PMID 40187738